CLINICAL TRIAL: NCT01973452
Title: A Double-Masked Placebo Controlled Clinical Trial of the Postoperative Opioid Sparing Effects of Intraoperative Dexmedetomidine Infusion for Thoracic Surgery
Brief Title: Placebo Controlled Clinical Trial of the Postoperative Opioid Sparing Effects of Intraoperative Dexmedetomidine Infusion for Thoracic Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-163
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2022-12

CONDITIONS: Pain
Keywords: Dexmedetomidine; Opioid; Thoracic Surgery
MeSH Terms: conditions — Pain | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Dexmedetomidine (Experimental): continuous infusion of 0.4 mcg/kg/hr
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): continuous infusion of 0.4 mcg/kg/hr
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine
  Arms: Dexmedetomidine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if the drug, Dexmedetomidine (also known as Precedex), can reduce pain for patients having Thoracic Surgery and therefore reduce the amount of opioid drug needed after surgery. It is a drug that is already approved by the FDA (Food & Drug Administration) for use as a sedative in hospitals and is currently used in the investigators Intensive Care Unit for this purpose. The investigators want to investigate if it also has pain relieving properties.

DETAILED DESCRIPTION:
The study involves the use of dexmedetomidine infusion intraoperatively during thoracic surgical procedures (not using an epidural) with discontinuation in the immediate postoperative period. A key feature in this study is to employ the drug infusion intraoperatively only.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ( ≥ 21 years old) scheduled for Thoracic Surgery

Exclusion Criteria:

* 2nd or 3rd degree heart block as assessed by preoperative EKG
* Use of dexmedetomidine within 28 days prior to day of surgery
* Use of long acting opioids pre-operatively 28 days prior to day of surgery
* Current or past diagnosis of a Major Psychiatric disorder precluding adequate outcome responses such as Schizophrenia, dementia, delirium etc. as recorded in the Pre-Operative Record.
* Documentation of congestive heart failure and Ejection fraction < 30% if recorded in the Pre-Operative Record.
* Planned use of an epidural for surgery or post-operative pain relief
* Contraindication to use of NSAID, Acetaminophen or IV opioids.
* Any known hypersensitivity to dexmedetomidine
* Pregnant or breastfeeding
* Abnormal liver function tests as related to the MSK guidelines for use of IV Acetaminophen

Yes or NO?; Is ALT greater than 2 x Upper Limit of Normal (> 75 U/L)?

* Abnormal renal function tests as related to contraindications to use of IV Ketorolac

Yes or No?; Is Serum Creatinine < 1.5 mg/dl?

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessia Pedoto, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center 1275 York Avenue, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexmedetomidine: continuous infusion of 0.4 mcg/kg/hr
  Dexmedetomidine
- Placebo: continuous infusion of 0.4 mcg/kg/hr
  Placebo
Period: Overall Study
Arm/Group | Dexmedetomidine | Placebo
Started | 165 | 166
Completed | 148 | 152
Not Completed | 17 | 14
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 10 | 9
Not completed — Ineligible | 1 | 1
Not completed — Surgery canceled by participant | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine | Placebo | Total
Number analyzed (Participants) | 148 | 152 | 300
Age, Continuous [Median (Full Range); unit: years] | 66 [57 to 71] | 65 [59 to 71] | 66 [57 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 64 | 130
  Male | 82 | 88 | 170
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 144 | 152 | 296
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 4 | 15
  White | 123 | 136 | 259
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 14 | 12 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 148 | 152 | 300

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Administered
Description: total opioid equivalents used postoperatively as measured by the total opioid administered in approximately the first 4 hours
Time Frame: up to 4 hours
Measure: Median (Full Range); unit: Morphine Milligram Equivalents
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 148 | 152
Morphine Milligram Equivalents | 4.0 [0.0 to 12.0] | 6.0 [0.0 to 14.0]

2. Secondary Outcome: Improves Analgesia
Description: as measured by change in Pain Numerical Rating Scale (NRS) preoperatively to postoperatively at rest and with activity (such as coughing). In the Pain Numerical Rating Scale (NRS), patients are asked to circle the number between 0 and 10 that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'
Time Frame: up to 24 hours
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 148 | 152
score on a scale | 4.0 [2.7 to 5.0] | 4.0 [2.8 to 5.0]

3. Secondary Outcome: Number of Participants With Episodes of Nausea or Antiemetic Doses and/or Sedation
Description: as measured by incidence of recorded nausea or the use of antiemetics and RASS sedation scores, respectively.
Time Frame: up to 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 148 | 152
Participants
  Participants with recorded nausea | 113 | 110
  Participants without recorded nausea | 35 | 42

ADVERSE EVENTS:
Time Frame: Up to 24 hours
Arm/Group | Dexmedetomidine | Placebo
All-Cause Mortality (participants affected / at risk) | 33/148 | 37/152
Serious Adverse Events (participants affected / at risk) | 5/148 | 8/152
Other Adverse Events (participants affected / at risk) | 0/148 | 0/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexmedetomidine (N=148) | Placebo (N=152)
Fever (General disorders) | 2 | 0
Lung infection (Infections and infestations) | 0 | 2
Intraoperative splenic injury (Injury, poisoning and procedural complications) | 0 | 1
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT01973452/Prot_SAP_000.pdf